CLINICAL TRIAL: NCT03215368
Title: A Population-Based Prospective Cohort Study to Examine the Effects of Maternal Pregnancy Exposure on Adverse Pregnancy Outcomes, Child Health and Their Development.
Brief Title: The Ma'Anshan Birth Cohort (MABC)
Status: Active, not recruiting | Type: Observational
Sponsor: Anhui Medical University (Other)
Collaborators: Ma'anshan Maternal and Child Health Care Hospital (Unknown)
Responsible Party: Principal Investigator, Fangbiao Tao, Principal Investigator, Anhui Medical University
Other Study IDs: 20131195
Record Dates: First submitted 2017-07-06; First posted 2017-07-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Environmental Exposure; Pregnancy Outcome; Birth Defects; Child Development; Maternal and Child Health; Health Problems in Pregnancy
Keywords: birth cohort study; environmental exposures; birth defects; pregnant outcomes; children development; Maternal and child health
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pregnancy and delivery：maternal blood, urine, cord blood and placenta. During infancy: urine and blood. During school age：Blood, urine and hair mother-child pairs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Ma'anshan Birth Cohort (MABC) is a population-based prospective pregnancy and birth cohort study that aims to explore the early environmental and genetic determinants of maternal and child health, with a focus on health outcomes including maternal health, children's cognitive and behavioral development, growth and physical development, video-screen behaviors, and asthma and allergic diseases.

MABC was officially launched in May 2013 at the Ma'anshan Maternal and Child Health Hospital in Anhui Province, and a total of 3,474 families were recruited as of September 2014 to continuously track the health status of mother-child pairs during pregnancy, delivery, and childhood, including basic family demographics, maternal pregnancy and birth history and past history, history of exposure to hazardous factors during pregnancy, children's diets and lifestyles, and children's physical and cognitive-behavioral development, MABC quantifies the attributional relationship between environmental chemicals, diet and nutrition, drug safety, psychological stress, lifestyle, biorhythm, endocrine metabolism and adverse birth outcomes, birth defects, neurodevelopmental disorders, developmental disabilities, etc., and identifies environmental, behavioral and genetic causative factors for birth defects and common developmental disorders, and identifies early warning signs and symptoms for early detection of birth defects. genetic causative factors, identify clinical biomarkers with early predictive effects, integrate and form a precise risk evaluation and early warning model, carry out regional comprehensive prevention and treatment applications, and promote the improvement of the quality of the birth population. Currently, MABC is conducting its 20th school-age follow-up visit.

ELIGIBILITY:
Inclusion Criteria

1. Permanent residents of Ma'anshan city;
2. Obstetric examination and delivery at Ma'anshan Maternal and Child Health Hospital;
3. Mother's age ≥ 18 years old and gestational week ≤ 14 weeks;
4. No serious neuropsychiatric disorders, with sufficient understanding and expression to complete the survey.

Exclusion criteria:

1. Intellectual disability or other serious mental disorders;
2. Suffering from serious underlying diseases and may have a significant impact on pregnancy outcome;
3. Those with poor compliance and difficulty in follow-up.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: From May 2013 to September 2014, 3474 pregnant women who first established a maternal health handbook in Ma'anshan Maternal and Child Health Hospital (MCHH) and were willing to undergo regular obstetric checkups and deliveries in the hospital were selected for inclusion in the cohort.
Sampling Method: Non-Probability Sample
Enrollment: 3474 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants with pregnancy complications | At delivery
  Including gestational diabetes, gestational hypertension, anemia, and hypothyroidism during pregnancy.
  Diagnosis by medical personnel at clinics
Numbers of participants with adverse pregnancy outcomes | At delivery
  Including preterm birth, low birth weight, macrosomia, abortion, stillbirth, and birth defects.
  Hospital information system collection

SECONDARY OUTCOMES:
Weight in kilogram changes during childhood | At birth and age at 42 days, 3 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 3.5 years, 4 years, 4.5years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years, 11years and 12 years
  Measured by health professionals in the clinic.
Height in centimeter changes during childhood | At birth and age at 42 days, 3 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 3.5 years, 4 years, 4.5years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years, 11years and 12 years
  Measured by health professionals in the clinic.
Early Child development | Age at 6 months, 48 months and 54 months
  Measured by Ages&Stages Questionnaires (ASQ). There are 6 questions in each of 5 domains of development: communication, gross motor, fine motor, problem-solving skills, and adaptive skills. Each question is given a 10 (yes), 5 (sometimes), or 0 (not yet) score according to the parents' answers. The sum scores (range from 0 to 300) and scores for each domain (range from 0 to 60) are calculated. Chinese norms are available for each domain, and any domain screened <2 SDs below the mean is considered a positive screening. A higher ASQ score means better development.
Child Psychological and Behavioural Development | Age at 48 months, 60 months and 72 months
  Measured by Strengths and Difficulties Questionnaire(SDQ). SDQ consisted of 25 entries scored on a 3-point scale from 0 to 2. 0: "Doesn't meet"; 1: "Somewhat meets"; 2: "Completely meets"; and the results were summarized into 5 factors: emotional factor, conduct factor, hyperactivity factor, peer factor, and pro-social factor, each with a score range of 0 to 10. The results were categorized into five factors: Emotional, Conduct, Hyperactivity, Peer, and Pro-social, each of which has a score range of 0-10 points. The sum of the scores of the first four factors is the total difficulty score of the SDQ, and the higher the score, the more serious the objective difficulty is. The higher the score, the better the pro-social ability.
Child Intelligence quotient | At age of 54 months
  Assessed by using Wechsler Preschool and Primary Scale of Intelligence-Fourth Edition-Chinese (WPPSI-IV（CN）), which can generate a full scale intelligence quotient score and five primary index scores including verbal comprehension, visual spatial, fluid reasoning, working memory, and processing speed. Intelligence quotient ranges from 40 to 160, in which less than 70 is defined as mental retardation
Child Sexual Development Indicators | At ages of 9-15 years for boys, and 8-14 years for girls
  Secondary sexual characters, Sexual hormones. Staging of puberty using Tanners classification: Testicular size of boys assessed by Prader's testerometer suggests possible precocious puberty if testicular development occurs before the age of 9 years in boys, and if breast development occurs before the age of 7.5 years or first menstruation occurs before the age of 10 years in girls. In order to further determine the existence and classification of precocious puberty, ultrasound examination of the uterus and ovaries for girls and ultrasound examination of the testes for boys are required. In addition to the above tests, bone age assessment, bone density test, adrenal gland ultrasound, thyroid function, sex hormone 6, alpha-fetoprotein measurement, growth hormone stimulation test and gonadotropin-releasing hormone stimulation test are also performed to further confirm the diagnosis.
Incidence of child overweight and obesity | At birth and age at 42 days, 3 months, 6 months, 9 months, 1 year, 1.5 years, 2 years, 2.5 years, 3 years, 3.5 years, 4 years, 4.5years, 5 years, 6 years, 7 years, 8 years, 9 years, 10 years, 11years and 12 years
  Measured by health professionals in clinic.
Fetal Head Circumference | At delivery.
  Measured by health professionals in clinic with ultrasound.
Fetal Abdominal Circumference | At delivery.
  Measured by health professionals in clinic with ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Fangbiao Tao, Study Director — Anhui Medical University
Locations (1):
- Ma'anshan Maternal and Child Health Care Hospital, Ma’anshan, Anhui, China

IPD SHARING:
Plan to Share IPD: No